CLINICAL TRIAL: NCT01691755
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Study to Assess the Efficacy, Safety and Tolerability of Aleglitazar Monotherapy Compared With Placebo in Patients With Type 2 Diabetes Mellitus (T2D) Who Are Drug-Naïve to Anti-Hyperglycemic Therapy
Brief Title: A Study of Aleglitazar in Patients With Type 2 Diabetes Mellitus Who Have Not Previously Received Anti-Hyperglycemic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC28034
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- aleglitazar (Experimental)
  Interventions: Drug: aleglitazar

INTERVENTIONS:
Drug: Placebo — oral doses once a day for 26 weeks
  Arms: Placebo
Drug: aleglitazar — 150 mcg orally once a day for 26 weeks
  Arms: aleglitazar

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will assess the efficacy, safety and tolerability of aleglitazar monotherapy compared with placebo in patients with type 2 diabetes mellitus who have not previously received anti-hyperglycemic therapy. Patients will be randomized to receive oral doses of 150 mcg aleglitazar once daily or placebo. The anticipated time on study treatment is 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of diabetes mellitus, type 2 within 12 months prior to screening
* Patients who have not received a anti-hyperglycemic medication for at least 12 weeks prior to screening and for not longer than 3 consecutive months in the past
* HbA1c >/=7% and </=9.5% at screening or within 4 weeks prior to screening and at pre-randomization visit
* Fasting plasma glucose </=240 mg/dL at pre-randomization visit
* Agreement to maintain diet and exercise habits during the study

Exclusion Criteria:

* Patients with Type 1 diabetes mellitus, secondary diabetes, diabetes resulting from pancreatic injury, or acute metabolic diabetic complications within the past 6 months
* Any previous treatment with thiazolidinedione or a dual peroxisome proliferator activated receptor (PPAR) agonist
* Any body weight lowering or lipoprotein-modifying therapy within 12 weeks prior to screening (except stable dose of statin)
* Symptomatic congestive heart failure classified as New York Heart Association class II-IV at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin HbA1c | From baseline to week 26

SECONDARY OUTCOMES:
Change in lipid profile | From baseline to week 26
Change from baseline in fasting plasma glucose | From baseline to week 26
Responder rate as defined of hemoglobin A1c (HbAc1) <7.0% (<6.5%) | From baseline to week 26
Change from baseline in homeostatic index of insulin sensitivity (HOMA-IS) | From baseline to week 26
Change from baseline in homeostatic index of beta cell function (HOMA-BCF) | From baseline to week 26
Safety: incidence of adverse events | 30 weeks (26 weeks treatment and 4 weeks follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (23):
  - Chino, California
  - Los Angeles, California
  - Santa Ana, California
  - Thousand Oaks, California
  - Upland, California
  - West Hills, California
  - Boynton Beach, Florida
  - Cooper City, Florida
  - Coral Gables, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - City of Saint Peters, Missouri
  - Greensboro, North Carolina
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Scranton, Pennsylvania
  - Tipton, Pennsylvania
  - Greer, South Carolina
  - Knoxville, Tennessee
  - Spokane, Washington
- Mexico (10):
  - Aguascaliente
  - Cuernavaca
  - Culiacán
  - Durango
  - Guadalajara
  - Mexico City
  - Monterrey
  - Pachuca
  - Querétaro
  - Tampico

REFERENCES:
- [Derived] Henry RR, Buse JB, Wu H, Durrwell L, Mingrino R, Jaekel K, El Azzouzi B, Andjelkovic M, Herz M. Efficacy, safety and tolerability of aleglitazar in patients with type 2 diabetes: pooled findings from three randomized phase III trials. Diabetes Obes Metab. 2015 Jun;17(6):560-565. doi: 10.1111/dom.12455. Epub 2015 Apr 8. PMID 25728612